CLINICAL TRIAL: NCT06110390
Title: High-flow Nasal Oxygen Therapy to Prevent Extubation Failure in Adult Trauma Intensive Care Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MRC-01-18-470
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Intensive Care; Airway Extubation; Critical Care; Oxygen Therapy

STUDY DESIGN:
Intervention Model Description: Cohort study. Permuted-block randomization to one of three arms
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be unaware of the intervention. Data analysis performed independently to assess outcome variables
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Flow Nasal Oxygen (Experimental): HFNO device
  Interventions: Device: High flow nasal oxygen
- Non-invasive ventilation (Experimental): Non-invasive ventilation via tight-fitting facemask
  Interventions: Device: High flow nasal oxygen
- Standard Oxygen therapy (Active Comparator): Facemask oxygen is the default device used
  Interventions: Device: High flow nasal oxygen

INTERVENTIONS:
Device: High flow nasal oxygen — An interface applied to the nostrils allowing fresh gas flows of up to 60 liters per minute and inspired oxygen concentrations of up to an fiO2 of 1.0
  Other Names: High flow nasal oxygen therapy; High flow nasal cannula

SUMMARY:
A significant proportion of patients who are intubated for trauma-related injuries, will fail the extubation process. This means that, when the decision has been made to remove the endotracheal tube, a certain proportion of these patients will require the endotracheal tube to be re-inserted. Global estimates for the rates of re-intubation range from 5-15% of all patients who have had attempted extubation on Intensive Care Units. The exact figures for intubated victims of trauma are not available. Re-intubation is associated with increased intensive care and hospital length of stay, increased morbidity, and the physical risks to the patient inherent with the intubation process. There is also some evidence that the rates of tracheostomy are higher in patients who have failed extubation. A number of interventions have been developed to help prevent extubation failure. Non-invasive ventilation and high-flow nasal oxygen are routinely employed in practice. However, there have been no specific studies of these interventions in TICU patients. High-flow nasal oxygen therapy (HFNO) has emerged over the last decade as a viable adjunct in the management of patients suffering from, or at risk of, hypoxemic respiratory failure. Within the intensive care unit settings, HFNO has been studies in terms of preventing intubation, but it has been evaluated more often in terms of preventing extubation failure.

Our study aims to answer the question of whether HFNO is effective at preventing extubation failure in intubated and ventilated victims of traumatic injuries. Previous studies on the same subject, are not based on unequivocal, robust RCTs with low risk of bias. Our primary outcome measure is re-intubation rates and secondary outcome measures are CO2 accumulation rates, atelectasis rates, nutrition status within first 24 hours post extubation, and post - extubation rates of vomiting. Ours will be a prospective, randomized clinical control study. There will be three arms to the study: a control arm, and two intervention arms. Randomization will be done on a permuted block basis. The control arm will be patients receiving standard oxygen therapy, and the intervention arms will be either High Flow Nasal Oxygen Therapy or Non-invasive Ventilation via mask. We propose that, when compared with either face-mask O2, NIV (CPAP), HFNO administered continuously for 24 hours post extubation of trauma patients on ICU, will result in better patient-related outcomes.

DETAILED DESCRIPTION:
High-flow nasal oxygen therapy (HFNO) has emerged over the last decade as a viable adjunct in the management of patients suffering from, or at risk of, hypoxemic respiratory failure. The mechanisms of its therapeutic benefit are not precisely understood but are thought to include a small but significant continuous positive airway pressure effect, and in the context of critically ill patients, the use of HFNO has been studied for the prevention of intubation, or as an alternative to Noninvasive Ventilation (NIV) for the prevention of intubation, in Type I respiratory failure patients, mostly with COPD or Heart Failure. Within the intensive care unit itself, HFNO has been studies in terms of preventing intubation, but it has been evaluated more in terms of preventing extubation failure. However, there have been no specific studies in Trauma Intensive Care Unit (TICU) patients. Patients suffering with polytrauma, who survive to TICU admission, are a unique population. There is a significant incidence of confusion and/or delirium post-extubation. In patients with respiratory failure post extubation, it is postulated (1) that the impaired mental state, however mild, may cause patients to a) be unable to tolerate NIV, b) swallow more air (on NIV) due to mild bulbar dysfunction, thus leading to an increased risk of regurgitation and possible aspiration pneumonitis. Furthermore, the use of NIV may c) impair effective oral nutrition in those patients without an NJ tube placed.

Re-intubation (failed extubation) is defined variably as the need to intubate a patient within 72 hours of extubation in the critical care unit. Re-intubation is associated with increased intensive care and hospital length of stay, increased morbidity, and the physical risks to the patient inherent with the intubation process. It is unclear which, if any, interventions can help reduce the rate of extubation failure in Trauma Intensive Care patients.

In this research study we are focusing on HFNO compared with NIV and conventional oxygen therapy in trauma patients to avoid reintubation.

We propose that, when compared with either face-mask oxygen, NIV (CPAP), HFNO administered continuously for 24 hours post extubation of trauma patients on ICU, will result in better patient-related outcomes.

Primary outcome measure:

Our primary outcome measure is re-intubation rate within 72 hours of extubation

Secondary outcome measures:

Our secondary outcomes measures are CO2 accumulation rates, atelectasis rates, nutrition status within first 24 hours post extubation, and post-extubation rates of vomiting.

Study design:

Prospective, randomized clinical control study. There will be three arms to the study: a control arm, and two intervention arms. Randomization will do on a permuted block basis. The control arm will be patients receiving standard oxygen therapy, and the intervention arms will be either High Flow Nasal Oxygen Therapy, or Non-invasive Ventilation via mask.

Study population:

All patients intubated on the Trauma Intensive Care Unit at Hamad General Hospital will be considered eligible for the study. Written informed consent will be obtained from next of kin (NOK) if available or by the treating physician as a surrogate if the NOK are not available. Study Population

Inclusion criteria: Adult intubated and ventilated patients who are victims of trauma and are being cared for on the Trauma Intensive Care Unit will be considered eligible for the study when they are considered fit for extubation.

Exclusion criteria:

* Patients who cannot be extubated (including patients requiring tracheostomy)
* Patients with cribriform plate fractures
* Patients with nasal occlusion for any reason
* Patients with unstable mid-face fractures

Sample size estimation:

Based on an anticipated improvement rate of 25% reduction in extubation failure (from 8% to 6%), using High-flow nasal Oxygen Therapy and NIV (CPAP) with margin of error of 5%, and confidence level of 95%, a total of 100 intubated trauma patients needs to be included in the study (50 for each group). Moreover, 50 patients with facemask O2 will be included as a comparative or control group.

The equation used for estimation of sample size:

The standard normal deviate for α = Zα = 1.960 The standard normal deviate for β = Zβ = 1.645 Pooled proportion = P = (q1*P1) + (q0*P0) = 0.103 A = Zα√P(1-P) (1/q1 + 1/q0) = 2.198 B = Zβ√P1(1-P1) (1/q1) + P0(1-P0) (1/q0) = 2.878 C = (P1-P0)2 = 0.292 Total group size = N = (A+B)2/C = 88 Continuity correction (added to N for Group 0) = CC = 1/ (q1 * |P1-P0|) = 23 So, a total of 113 cases are required for this study (38 cases in each group), since the target reduction of extubation failure (effect size is small from 8% to 6% i.e., 25%) we prefer to include 50 cases in each group.

Allocation ratio: 1:1:1

Study procedures:

1. The enrollment for the study will begin once patient is ready for extubation and at the same time will be randomized to the study arms.
2. All intubated patients with next of kin /deferred consent will be enrolled
3. The respiratory therapist will apply the intervention type based on physician order

The study participants will be unblinded, as intervention is in the form of face mask O2, High flow nasal oxygen and NIV. These cannot be used in a blind approach.

We have developed a flow-chart for the study participants, which include an escalation pathway. If HFNO fails, patients are escalated to NIV- CPAP. If Facemask O2 fails, patients are escalated to HFNO or NIV, depending on treating clinician preference. The maximum observation time allowed to test whether intervention is effective is one hour. Re-intubation requirement will be assessed by treating clinician depending on ABG/oxygenation/CO2 or WOB criteria, or 'clinician-judgement'. This may occur at any time.

Screening and enrollment: The data will be prospectively collected for all intubated enrolled patients admitted to the Hamad General Hospital trauma ICU between 1 October 2020 and 31 December 2023.

all ventilated patients will be recruited based on next of kin/deferred consent during the study period for the study in trauma ICU. The enrollment of the patients will be for 3 years from start of study period

Follow up: Each patient will be followed up for 72 hours post extubation as a part of study

Informed Consent:

Unconscious patients with severe injury will not be able to provide informed consent. This trial will therefore use "Exception from Informed Consent Requirements for Emergency Research" (Policy # RES 11026) which involves the most vulnerable population of study subjects (i.e., a population with no capacity to control what happens to them and no capacity to consent, where the emergency circumstances require prompt action and generally provide insufficient time and opportunity to locate and obtain consent from each subject's family member).

Every possible effort will made to contact the subject's family member to obtain consent. However, it may be difficult to contact family members of migrant workers within the initial time frame in the emergency department. In such situation, initially the deferred consent document will be signed by two privileged physicians, one of whom will be the treating physician. After regaining complete consciousness patient will be asked for continuation in the study and if the subject agrees written informed consent will be obtained.

As soon as is reasonably possible and appropriate the patient's NOK/person responsible will be informed of the patient's inclusion in the research and will be informed of the option to withdraw the patient from it without any reduction in quality of care. If the NOK/person responsibly chooses to withdraw their consent for continued participation, they will be asked for permission to use the data collected up to that time.

Patients who recover sufficient cognition to understand the explanation of the study will be asked to consent to continue in the study or be offered the chance to withdraw. If the patient chooses to withdraw from the study, they will be asked for permission to use their data up to the time of withdrawal.

All interaction between research staff and participants and their relatives will take into consideration the stress or emotional factors associated with critical illness and ensure that the dependency of potential participants and their relatives on medical personnel providing treatment does not compromise their actual or perceived freedom of decision making to participate.

Risk This study does not add any novel risks to patients as all the interventions are currently used as part of standard bundles of care. Potential complications include local trauma, discomfort and pressure areas, epistaxis and gastric distension from the use of NIV. Dry airways are a potential complication of both face mask O2 and HFNCO2. These risks are the same as if the patients are receiving a standard clinical care of treatment or not participating in the research

Data Collection & Integrity:

The data will be prospectively collected for all intubated enrolled patients admitted to the Hamad General Hospital trauma ICU from 1 October 2020 to 31 December 2023. Patient data includes Age, Gender, Mechanism of injury, associated injury, Date & time of Trauma, arrival to Trauma room, admission, Vital signs in Trauma ICU, GCS, intubation date, and injuries, duration of hospital, ICU stay and mortality.

Most importantly, the group allocation will be to Facemask O2, NIV-CPAP, or HFNO. We will compare the rates of re-intubation using a p-value of < 0.05 to confirm a statistical difference.

Data will be anonymously collected, and the data sheet will be secured with the principal investigator. The name of the patients will not be disclosed and kept confidential. The study is complying with the "Records-based study" profile that was described by corresponding section of the collaborative Intuitional Training Initiative (CITI). Patients' name and HC numbers will be used temporarily and only upon data collection and cleaning, to prevent duplication and allows proper re-access to the corresponding data to refine them. Both the name and HC number will be deleted immediately after data entry and coding.

Data will be presented as proportions, medians, or mean ± standard deviation (SD) as appropriate. Differences in categorical variables between respective groups will be analyzed using the chi square test. The continuous variables will be analyzed using Student's t-test. For skewed continuous data non-parametric Mann-Whitney test will be performed. Two-tailed P values of <0.05 will be considered significant. Data analysis will be carried out using the Statistical Package for Social Sciences version 18 (SPSS Inc. USA).

Quality Assurance, Monitoring & Safety:

The research team will be responsible for the data collection, entry, confidentiality and maintaining the quality of the data. It will also oversee the ethical conduct of the trial, safety, protection, privacy and confidentiality of the subjects and adherence to the study protocol. We will follow the instructions from institutional review committee to setup any independent monitoring committee, if needed.

ELIGIBILITY:
Inclusion Criteria:

* Adult intubated and ventilated patients who are victims of trauma and are being cared for on the Trauma Intensive Care Unit will be considered eligible for the study when they are considered fit for extubation.

Exclusion Criteria:

* Patients who cannot be extubated (including patients requiring tracheostomy)
* Patients with cribriform plate fractures
* Patients with nasal occlusion for any reason
* Patients with unstable mid-face fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2020-10-17 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Reintubation rate | 72 hours
  How many patients who have experienced extubation require re-intubation.

SECONDARY OUTCOMES:
Nutritional intake achieved | 24 hours post extubation
  Estimated caloric intake
Post extubation rates of vomiting | 24 hours
  How many patients vomited post extubation
Amount of carbon dioxide retention | 24 hours post extubation
  Surrogate marker for insufficient ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Rizoli, Study Chair — Hamad Medical Corporation
Locations (1):
- Hamad General Hospital, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
Physiological data including arterial blood gas results may be shared in future